CLINICAL TRIAL: NCT02696252
Title: Comparison of G5® Mobile Continuous Glucose Monitoring System Accuracy When Using an Automated Applicator vs. a Manual Sensor Applicator
Brief Title: G5® Mobile Continuous Glucose Monitoring System Automated vs. Manual Sensor Applicator
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-901800
Record Dates: First submitted 2016-01-25; First posted 2016-03-02 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus
Keywords: Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases
MeSH Terms: conditions — Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CGM Users

SUMMARY:
Comparison of G5® Mobile Continuous Glucose Monitoring System Accuracy When Using an Automated Applicator vs. a Manual Sensor Applicator

DETAILED DESCRIPTION:
The objective of the study is to demonstrate the performance, i.e. efficacy of the G5x System with the automated applicator is no worse than that of the commercial Dexcom G4 TM PLATINUM Continuous Glucose Monitoring System (G4 System) with the manual applicator.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 or older
* Diagnosis of Type 1 diabetes or Type 2 diabetes
* Willing to participate in a clinic session involving venous sampling for evaluation of study end point

Exclusion Criteria:

* Use of acetaminophen
* Known allergy to medical-grade adhesives
* Pregnancy
* Hematocrit outside specification of the study-assigned blood glucose meter

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and pediatrics with diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
proportion of blood glucose values, compared between CGM and a lab glucose analyzer that are matched relative to a diabetes accuracy measurement of %20/20 mg/dL | 7 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - AMCR Institute, Escondido, California
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Joslin Diabetes Center, Boston, Massachusetts
  - Clinical Trials of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided